CLINICAL TRIAL: NCT01080105
Title: Technology Assisted Behavioral Intervention for the Prevention of Depression
Brief Title: Internet Intervention for the Prevention of Depression - Approaches to Improving Mood
Acronym: AIM
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This is withdrawn because we started working on studies that are funded.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NU IRB STU00020637
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Individuals at Risk for Depression
Keywords: Depression Prevention; Prevention; Major Depressive Disorder; Internet; Technology Assisted
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AIM + surveillance (Experimental): Participants will receive access to the AIM website and calls from a motivational coach for 12 weeks plus an additional year of surveillance and optional coach support.
  Interventions: Behavioral: AIM Web based intervention + surveillance
- AIM intervention (Experimental): Participants will receive access to the AIM web based intervention and calls from a motivational coach for 12 weeks
  Interventions: Behavioral: AIM web based intervention
- Educational website (Active Comparator): Participants will be given access to a static website with depression prevention related materials and handouts.
  Interventions: Behavioral: Educational website

INTERVENTIONS:
Behavioral: AIM Web based intervention + surveillance — The web based intervention will include 12 weeks of Internet-based cognitive behavioral therapy combined with brief telephone and email support from a coach. Surveillance will consist of monthly screening of depression symptoms and outreach from the coach should there be an increase in symptoms.
  Arms: AIM + surveillance
Behavioral: AIM web based intervention — The web based intervention will include 12 weeks of Internet-based cognitive behavioral therapy combined with brief telephone and email support from a coach.
  Arms: AIM intervention
Behavioral: Educational website — Participants will receive access to a static educational website for 12 weeks.
  Arms: Educational website

SUMMARY:
This study will develop and evaluate the effectiveness of a technology-assisted behavioral intervention, consisting of Internet-based cognitive behavioral therapy combined with telephone and email support, in preventing depressive symptoms and improving treatment adherence in individuals at risk of major depressive disorder.

DETAILED DESCRIPTION:
Depression is common, with one-year prevalence rates of major depressive disorder (MDD) estimated to be between 6.6-10.3% in the general population. Depression imposes a very high societal burden in terms of cost, morbidity, suffering, and mortality. Yet only about 20% of all patients referred for psychotherapy ever enter treatment, and of those who initiate treatment, nearly half drop out before completion. Given the limitations of treatment and the significant burden of depression, research into the prevention of depression is needed. There is a dearth of research related to the effective prevention of depression.

Delivering an intervention through telecommunication technologies, such as the telephone and Internet, has the potential to overcome many of the barriers to existing depression prevention interventions. For example, telephone- and Web-based interventions can reduce cost, extend specialized treatment over broad geographic areas, and permit considerable flexibility in scheduling of treatment components. Approaches to Improving Mood (AIM) is a specific form of a telecommunication behavioral intervention that incorporates Web-based Internet, e-mail, and telephone intervention. Further study is needed to determine the effectiveness of AIM in preventing depressive symptoms and improving attrition from treatment rates in people at risk for MDD. The study will compare the effectiveness of the AIM program with a one year surveillance follow up with the effectiveness of the AIM program alone and a website offering information on depression prevention in preventing depressive symptoms and improving treatment adherence in individuals at risk of MDD.

Participation in the treatment phase of this study will last 12 weeks. All participants will first undergo initial assessments that will include a telephone interview and a series of questionnaires about mood. Eligible participants will then be assigned randomly to receive AIM + surveillance, AIM alone, or the education website. All participants will undergo 12 weeks of a Web-based Internet intervention consisting of modules to help them learn skills to manage their moods. Participants will be asked to access the Web site every day or two to complete the modules and to practice the learned techniques. Participants assigned to AIM + surveillance and AIM alone will also receive a weekly telephone-based motivational intervention from a coach and will be able to communicate with the coach via email throughout the first 12 weeks of treatment. Participants assigned to the education group will be given access to a website but no assistance from a coach. All participants will undergo repeat initial assessments at Weeks 6, 12 (end of treatment) and at 3 months, 6 months, 9 months and 12 months following the completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* PredictD Risk Score of .130
* Has a telephone, e-mail account, computer, and broadband access to the Internet.
* Is able to speak and read English.
* Is at least 19 years of age.
* Is able to give informed consent.

Exclusion Criteria:

* Has DSM-IV diagnosis of Major Depressive Episode assessed using the MINI
* Has hearing or voice impairment that would prevent participation in psychotherapy.
* Has visual impairment that would prevent use of the workbook and completion of assessment materials.
* Meets criteria for dementia by scoring < 25 on the Telephone Interview for Cognitive Status (TICS).
* Is diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, current post-traumatic stress disorder (PTSD), current substance abuse, or other diagnosis for which participation in a clinical trial of psychotherapy may be either inappropriate or dangerous. Patients with substance abuse diagnoses who have been clean and sober for 3 months will be admitted if otherwise eligible.
* Is currently receiving individual psychotherapy or planning to receive psychotherapy during the 12-week treatment phase of the study.
* Is planning to be out of town or unavailable for treatment for 4 weeks or more during the scheduled treatment time.
* Exhibits severe suicidality, including ideation, plan, and intent.
* Has initiated treatment with an antidepressant in past 10 days. Once patients have been on a stable dose for 10 days and do not have an appointment with a physician or psychiatrist to change this dose, the patient will be eligible based on this criterion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Depression, as assessed by Quick Inventory of Depressive Symptoms (QIDS), the Patient Health Questionnaire-9 (PHQ-9), and the Mini International Neuropsychiatric Interview (MINI) Disorders-Major Depressive Disorders Module | Measured at baseline, week 6, week 12 and month 3, month 6, month 9 and month 12
Website utilization (e.g., number of logins, average visit length, total time spent on the site, number of exercises completed), Attrition and cost effectiveness. | From baseline through 12 month follow-up

SECONDARY OUTCOMES:
Anxiety, impact on work, social support | Measured at baseline, week 6, week 12 and month 3, month 6, month 9 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mohr, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States